CLINICAL TRIAL: NCT05750797
Title: The Nationwide Real-world Status of Oral Corticosteroid Use in Patients With Asthma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Joon Young Choi (Other)
Collaborators: Seoul St. Mary's Hospital (Other); Hallym University Medical Center (Other); Konkuk University Hospital (Other)
Responsible Party: Sponsor-Investigator, Joon Young Choi, Clinical assistant professor, Incheon St.Mary's Hospital
Organization: Incheon St.Mary's Hospital (Other)
Other Study IDs: ESR-21-21329
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Asthma; Corticosteroid
MeSH Terms: conditions — Asthma | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Oral corticosteroids — The prescription of OCS will be analyzed. OCS included betamethasone, deflazacort, dexamethasone, hydrocortisone, methylprednisolone, prednisolone, and triamcinolone.

SUMMARY:
The Health Insurance Review and Assessment Service (HIRA) database contains nationwide claim data. By utilizing this database, the investigators aimed to analyze the current status of OCS use in South Korea by using HIRA database.

DETAILED DESCRIPTION:
South Korea has a compulsory universal health insurance system for entire Korean population. The number of people who are covered was more than 50 million. The Health Insurance Review and Assessment Service (HIRA) database contains nationwide claim data. By utilizing this database, the investigators have performed many studies regarding asthma in South Korea. In this study, the investigators aimed to analyze the current status of OCS use in South Korea by using HIRA database.

Primary outcome was the OCS prescription in all patients with asthma. Secondary outcome was OCS prescription according to the asthma severity, age, sex, socioeconomic status and the type of hospital.

Inclusion criteria was 1) Age ≥ 15 years; 2) ICD-10 codes for asthma (J45.x-J46) as the primary or within fourth secondary diagnosis; 3) use of more than one drug for asthma at least twice per year (long acting muscarinic antagonist (LAMA), long acting beta2 agonist (LABA), ICS, ICS+LABA, short acting muscarinic antagonist (SAMA), short acting beta2 agonist (SABA), SAMA+SABA, theophylline, leukotriene antagonist, systemic corticosteroids, or systemic beta agonist).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 15 years;
* ICD-10 codes for asthma (J45.x-J46) as the primary or within fourth secondary diagnosis
* use of more than one drug for asthma at least twice per year (long acting muscarinic antagonist (LAMA), long acting beta2 agonist (LABA), ICS, ICS+LABA, short acting muscarinic antagonist (SAMA), short acting beta2 agonist (SABA), SAMA+SABA, theophylline, leukotriene antagonist, systemic corticosteroids, or systemic beta agonist).

Exclusion Criteria:

• Those who are not in the insurance system

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those who were diagnosed and treated as Asthma from 1-Jan-2019 to 31-Dec-2019
Sampling Method: Non-Probability Sample
Enrollment: 800000 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
OCS prescription rates | 1-year
  Analysis the OCS prescription in all patients with asthma

SECONDARY OUTCOMES:
OCS prescription according to the asthma severity | 1-year
OCS prescription according to age | 1-year
OCS prescription according to sex | 1-year
OCS prescription according to socioeconomic status | 1-year
OCS prescription according to the type of hospital | 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St. Mary's Hospital, Incheon, Gyeongki, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD cannot be publicaly available due to restriction.